CLINICAL TRIAL: NCT03879811
Title: Phase II Study of Temozolomide and Nivolumab in MMR-Proficient Colorectal Cancer (CA209-8JN)
Brief Title: Determining the Effects of Temozolomide Followed by Nivolumab in Patients With Colorectal Cancer
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No accrual
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-545
Record Dates: First submitted 2019-03-15; First posted 2019-03-19 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2019-12

CONDITIONS: Colorectal Cancer
Keywords: MMR-Proficient Colorectal Cancer; Temozolomide; Nivolumab; Memorial Sloan Kettering Cancer Center; 18-545
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Nivolumab

STUDY DESIGN:
Intervention Model Description: Simon two-stage design, single arm study
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MMR-Proficient Colorectal Cancer (Experimental): The first 3 subjects will receive oral TMZ at 150mg/m2 day 1 to 5 during cycle
  1, followed by nivolumab via IV infusion at 480 mg every four weeks (Q4W) starting 4 weeks after TMZ day 1 (i.e. Cycle 2 day 1). Nivolumab will continue for up for 2 years maximum. If confirmed that TMB increased in at least 2 of 3 subjects following 1 cycle of TMZ, then subsequent patients will continue to receive TMZ during cycle 1 only, and the original three participants will not be replaced. If it is determined that TMB did not increase following 1 cycle of TMZ, then subsequent patients will receive TMZ up to cycle 3, those first 3 patients will discontinue further Nivolumab and be replaced and an additional 6 patients will initially be enrolled. If confirmed that TMB increased in at least 1 of 6 subjects following 3 cycles of TMZ, then 12 more patients will be allowed to enroll for a total of 18 in stage I.
  Interventions: Drug: TMZ; Drug: Nivolumab

INTERVENTIONS:
Drug: TMZ — Oral TMZ at 150mg/m2
Drug: Nivolumab — Nivolumab via IV infusion at 480 mg every four weeks (Q4W) starting 4 weeks after TMZ day 1

SUMMARY:
The purpose of this study is to find out whether temozolomide followed by nivolumab is an effective treatment for MMR-proficient colorectal cancer, while causing few or mild side effects.

ELIGIBILITY:
Inclusion Criteria:

* Subject or legally authorized representative, is willing and able to provide written informed consent/assent for the trial
* Histologically- or cytologically- confirmed CRC
* Locally advanced or metastatic CRC
* Confirmation of MGMT promoter methylation on archived tissue by PCR analysis (any time).
* MGMT promoter methylation is determined using the ARUP laboratory assay (or similar). Total methylation is calculated as an average across listed CpG sites. Total methylation of 0-9 percent is reported as "Not detected" 10-29 percent as "Low level" and equal or more than 30 percent as "Detected". Patients will require MGMT promoter methylation to be "detected" in order to be eligible.
* Undergone testing for MSI/dMMR and determined to be MSS or MMR proficient
* Subjects must be refractory or intolerant to at least 2 lines of standard chemotherapy, according to NCCN guidelines for patients eligible for intensive therapy. At a minimum, such therapies should include regimens containing oxaliplatin or irinotecan in combination with a fluoropyrimidine (e.g., FOLFOX or FOLFIRI or their variants).
* At least one index lesion which is measurable based on RECIST 1.1
* Be >/= 18 years of age on day of signing informed consent
* Consent for tumor biopsies and blood draws for research purposes
* Have an ECOG performance status of 0 or 1
* Demonstrate adequate organ function as defined in Table 6.1, all screening labs should be performed within 28 days of treatment initiation.

Adequate Organ Function Laboratory Values

Hematological

* Absolute neutrophil count (ANC) >/= 1,500/mcl
* Platelets >/= 100,000/mcl
* WBC >/= 2000/ul
* Hemoglobin >/= 9.0 g/dL

Renal

* Serum creatinine </= 1.5 x upper limit of normal (ULN) OR
* Measured or calculated creatinine clearance (GFR can also be used in place of creatinine of CrCl) >/= 60 mL/min for subject with creatinine levels > 1.5 x institutional ULN (Creatinine clearance should be calculated per institutional standard)

Hepatic

* Serum total bilirubin </= 1.5 x ULN -OR- Direct bilirubin </= ULN for subjects with total bilirubin levels > 1.5 ULN
* AST (SGOT) and ALT (SGPT) </= 2.5 x ULN -OR- </= 5 x ULN for subjects with liver metastases
* Female subject of childbearing potential should have a negative serum pregnancy within 2 weeks prior to starting treatment
* Female subjects of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity for the course of the study through 5 months after the last dose of study medication. Subjects of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
* Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 7 months after the last dose of study therapy (defined in section 7.1). In addition, male subjects must be willing to refrain from sperm donation during this time.

Coagulation

* International Normalized Ratio (INR) or Prothrombin Time (PT) </= 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants
* Activated Partial Thromboplastin Time (aPTT) </= 1.5 x ULN unless subject is receiving anticoagulant therapy as long as PT or PTT is within therapeutic range of intended use of anticoagulants

Exclusion Criteria:

* Subject is currently participating in or has participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (>10 mg/day prednisone, or equivalent) or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment. inhaled or topical steroids are permitted in the absence of active autoimmune disease
* Prior chemotherapy, targeted small molecule therapy, or biological therapy, within 2 weeks prior to study Day 1 or who has not recovered (i.e., </= Grade 1 or at baseline) from adverse events due to a previously administered agent (exc. alopecia)
* If subject received major surgery, they must have recovered adequately prior to starting therapy
* Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis. Subjects with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least four weeks prior to the first dose of trial treatment any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment,
* Has an active, known or suspected autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy, type 1 diabetes mellitus are permitted. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Subjects with hypothyroidism stable on hormone replacement or Sjorgen's syndrome will not be excluded from the study.
* Has evidence of known interstitial lung disease or active, non-infectious pneumonitis
* Has an active infection requiring systemic therapy
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the subject's participation for the full duration of the trial, or it is not in the best interest of the subject to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-screening or screening visit through 5 months for females, 7 months for males after the last dose of trial treatment
* Prior anti-PD-1, anti-PDL-1, anti-PDL-2, anti-Cytotixic T-lymphocyte-associated antigen-4 (CTLA-4) antibody or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways
* Has a known history of Human Immunodeficiency Virus (HIV) (HIV 1/2 antibodies)
* Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment
* Subjects is a prisoners or compulsory detained

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-03-13 (Actual); Primary Completion 2021-03 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
response rate of TMZ followed by nivolumab in participants with MMR-proficient Colorectal Cancer | up to 2 years
  Response determined by RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Neil H Segal, MD, PhD, Principal Investigator — Memorial Sloan Kettering Cancer Center

IPD SHARING:
Plan to Share IPD: Yes
Here is the final approved MSK data sharing statement for posting on any trial opened 1/1/19 or later -
  • Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Related Info — http://www.mskcc.org